CLINICAL TRIAL: NCT04219410
Title: Assessment of a Modified Minimally Invasive Esophagectomy
Status: Completed | Type: Observational
Sponsor: Kaiser Permanente (Other)
Responsible Party: Principal Investigator, Andy Avins, Senior Research Scientist, Kaiser Permanente
Other Study IDs: 1279152-4
Record Dates: First submitted 2020-01-03; First posted 2020-01-07 (Actual); Last update posted 2020-01-07 (Actual); Status verified 2020-01

CONDITIONS: Esophageal Cancer
MeSH Terms: conditions — Esophageal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cases: Patients who underwent minimally invasive esophagectomy with this novel procedure at Kaiser Permanente, Northern California, Oakland Medical Center
  Interventions: Procedure: Fully minimally invasive esophagectomy

INTERVENTIONS:
Procedure: Fully minimally invasive esophagectomy — Esophagectomy using a novel fully minimally invasive approach

SUMMARY:
This is a retrospective case series of a novel fully minimally invasive esophagectomy procedure for patients with primary esophageal cancer.

ELIGIBILITY:
Inclusion Criteria:

* patient with primary esophageal cancer of any cell type
* underwent the novel minimally invasive esophagectomy procedure at the Kaiser Permanente Northern California Oakland Medical Center by one of the study author-surgeons

Exclusion Criteria:

* non-elective procedure
* less than 90 days of post-discharge follow-up

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive sample of all patients undergoing the novel minimally invasive esophagectomy procedure at the Kaiser Permanente Northern California Oakland Medical Center during the study period
Sampling Method: Non-Probability Sample
Enrollment: 142 (Actual)
Dates: Start 2013-01-01 (Actual); Primary Completion 2016-08-31 (Actual); Study Completion 2016-08-31 (Actual)

PRIMARY OUTCOMES:
Hospital length of stay | Through study completion, an average of 2.9 years
  Hospital length of stay

SECONDARY OUTCOMES:
Intensive care unit length of stay | Through study completion, an average of 2.9 years
  Intensive care unit length of stay
Feeding tube placement | Intra-operatively
  Feeding tube placement
Number of patients with inpatient mortality | Through study completion, an average of 2.9 years
  Number of patients with inpatient mortality
90-day total mortality | 90 days post discharge
  90-day total mortality
Number of patients with hospital readmission within 30 days | 30 days post discharge
  Number of patients with hospital readmission within 30 days
Number of patients with complications | Hospital stay and 30 days post discharge
  Number of patients with medical and surgical complications both inpatient and post-discharge

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Avins, MD, MPH, Principal Investigator — Kaiser Permanente

IPD SHARING:
Plan to Share IPD: No